CLINICAL TRIAL: NCT06423833
Title: Trendelenburg Maneuver Versus Passive Leg Raising Test for Fluid Responsiveness in High-Risk Surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Fatma Mohamed Samy Elaiashy, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 36264MD32/2/23
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Trendelenburg Maneuver; Passive Leg Raising; High-Risk Surgical Patients

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trendelenburg maneuver (Experimental): The investigator will measure changes in velocity time integral (VTI) and stroke volume (SV) during Trendelenburg maneuver (TM) in high-risk surgical patients by trans-thoracic Doppler echo cardiography
  Interventions: Diagnostic Test: Trendelenburg maneuver (TM)
- Passive leg raising test (Active Comparator): The investigator will measure changes in velocity time integral (VTI) and stroke volume (SV) during passive leg raising (PLR) test in high-risk surgical patients by trans-thoracic Doppler echo cardiography
  Interventions: Diagnostic Test: Passive leg raising test

INTERVENTIONS:
Diagnostic Test: Trendelenburg maneuver (TM) — The investigator will measure changes in velocity time integral (VTI) and stroke volume (SV) during Trendelenburg maneuver (TM) in high-risk surgical patients by trans-thoracic Doppler echo cardiography.
  Arms: Trendelenburg maneuver
Diagnostic Test: Passive leg raising test — The investigator will measure changes in velocity time integral (VTI) and stroke volume (SV) during Passive leg raising (PLR) test in high-risk surgical patients by trans-thoracic Doppler echo cardiography.
  Arms: Passive leg raising test

SUMMARY:
The aim of this study is to evaluate whether Trendelenburg maneuver can be used to predict fluid responsiveness in high-risk surgical patients in intensive care unit as compared to Passive Leg Raising test.

DETAILED DESCRIPTION:
Passive Leg Raising test is a well validated dynamic method to predict fluid responsiveness with many advantages as it doesn't use fluid loading, its effect is reversible, and it doesn't rely on heart-lung interaction. However, it has many limitations as (has false negative effect in patients with intra-abdominal hypertension), also, it may not be suitable in some surgical patients.

Trendelenburg maneuver (TM) is often used to treat hemodynamic unstable patients when hypovolemia is suspected, through a mechanism similar to Passive Leg Raising test Yonis, et al reports that change in cardiac output during Trendelenburg maneuver is a reliable predictor of fluid responsiveness in patients with acute respiratory distress syndrome in prone position under protective ventilation. Another study reports that change in velocity time integral during trendelenburg maneuver predicts fluid responsiveness in cardiac surgical patients in operating rooms

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old.
* Criteria of high-risk surgical patients:

  1. Elderly ≥ 70 years old undergoing major surgery.
  2. Physical status ≥ 3 or more undergoing major surgery.
  3. Major intraoperative hemorrhage with Surgical Apgar Score (SAS 0-4).
  4. Emergency of upper abdominal surgery.
* Criteria of hypoperfusion ≥ 2 or more the following:

  1. Mean arterial blood pressure < 65 mmHg.
  2. Urine output < 0.5 ml/Kg/hr.
  3. Capillary refilling time > 4 seconds.
  4. Blood lactate > 2 mmol/L.
  5. ScvO2 < 70%.
  6. CO2 gap > 6 mmHg.
* Provided that:SpO2 ≥ 90% and Hb ≥ 7 g/dl.

Exclusion Criteria:

* Patients with body mass index > 35 kg/m2.
* Pregnant female.
* Contraindications to the Trendelenburg position or PLR test (major head trauma, intra-abdominal hypertension and gastric retention).
* Poor echo window or unsatisfactory cardiac echogenicity (an inability to correctly align the Doppler beam to generate reliable velocity time integral measurements at the left ventricular outflow tract [LVOT]).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
The validity of Trendelenburg maneuver | At the end of Trendelenburg maneuver within 1 minute
  Measurement of the validity of Trendelenburg maneuver to predict fluid responsiveness by measuring the percentage change in velocity time integral (VTI) by Doppler echocardiography in high risk-surgical patients.

SECONDARY OUTCOMES:
Correlation between the accuracy of the percentage change in velocity time integral (VTI) during Trendelenburg maneuver and passive leg raising test (PLR) test | At the end of Trendelenburg maneuver and passive leg raising test within 1 minute
  Correlation between the accuracy of the percentage change in velocity time integral (VTI)during Trendelenburg maneuver and passive leg raising test will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author